CLINICAL TRIAL: NCT00212797
Title: Prospective, Double-Blind, Randomized, Placebo-Controlled Dose Finding Study of the Efficacy and Safety of 2 Target Doses of Org 34517 Used as Adjunctive Therapy in Subjects With Psychotic Major Depression (Major Depressive Episode, Severe, With Psychotic Features).
Brief Title: A Study to Determine the Efficacy and Safety of 2 Doses of Org 34517 as Adjunctive Therapy in Subjects With Psychotic Major Depression (28130)(P05845)
Acronym: Hermes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05845; Protocol 28130
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Depression; Depressive Disorders; Psychotic Disorders
MeSH Terms: conditions — Depression; Depressive Disorder; Psychotic Disorders | interventions — Org 34517

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Org 34517_1 (Experimental): low dose Org 34517
  Interventions: Drug: Org 34517
- Org 34517_2 (Experimental): high dose Org 34517
  Interventions: Drug: Org 34517
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Org 34517 — low dose Org 34517
  Arms: Org 34517_1
Drug: Org 34517 — high dose Org 34517
  Arms: Org 34517_2
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether subjects with psychotic major depression benefit from adjunctive treatment with Org 34517. Two doses of Org 34517 will be compared to placebo in this international multicenter study. The duration of this trial is 6 weeks.

DETAILED DESCRIPTION:
Major depression with psychotic features (psychotic depression) is the most debilitating disorder in the depressive disorders spectrum. It is associated with severe symptoms, prolonged course, poorer response rates, more residual symptoms, more frequent relapses and higher mortality, as compared to major depressive disorder.

The markedly abnormal HPA axis functioning in psychotic depression has encouraged research to investigate whether the HPA axis would be a target for pharmacotherapy in depression.

The primary purpose of this study is to determine whether subjects with psychotic major depression benefit from adjunctive treatment with GR antagonist Org 34517. Two doses of Org 34517 will be compared to placebo in this international multicenter study. The duration of this trial is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* have provided voluntary written informed consent for trial participation after the scope and nature of the investigation were explained to them, and before starting any trial-related activities (before Screening);
* be able to speak, read, understand, respond to questions, and follow

instructions in English or their native language;

* have DSM-IV severe depressive episode with psychotic features, as

diagnosed by the MINI for single or recurrent episodes (296.24 or 296.34);

have a score on PANSS item "Delusions" AND/OR "Hallucinatory behavior" of at least 4 at Screening and Baseline;

* have a PANSS Positive Scale score of at least 16 at Screening and Baseline;
* have a total score of at least 18 on the HAMD 17-item scale at Screening and Baseline;
* be on a stable dose of "usual treatment", which had to consist of an

antidepressant, an antipsychotic, a mood stabilizer or any combination of these 3 drug classes;

* be between 18 and 75 years of age (inclusive) at Screening;
* be willing to be hospitalized for at least 11 days from Screening onwards.

Exclusion Criteria:

* have any other current psychiatric diagnosis (according to the MINI) except MDD, such as organic mental syndromes and disorders, delirium or anxiety disorders;
* have a lifetime psychiatric diagnosis of psychotic disorders (according to the MINI), or a MINI diagnosis of past manic episode;
* be at significant risk of committing suicide, as indicated by a score greater than 9 on the revised InterSePT Scale for Suicidal Thinking (ISST);
* be currently treated with carbamazepine or valproate;
* be currently treated with midazolam;
* be treated with electroconvulsive therapy in the current episode;
* be currently treated with more than one antidepressant;
* be currently treated with more than one antipsychotic;
* be currently treated with more than one mood stabilizer;
* have a "usual treatment" started or discontinued in the 2 weeks before

Randomization;

* have a "usual treatment" dose change within the week prior to

Randomization;

* have any clinically unstable or uncontrollable renal, hepatic, respiratory,

hematological, cardiovascular or cerebrovascular disease that would put the patient at risk of safety or bias assessment of efficacy;

have known hypersensitivity reactions to glucocorticoid antagonists;

* have any clinically significant abnormal laboratory data (e.g. aspartate amino transferase (ASAT) and/or alanine amino transferase (ALAT) values > 2x normal range upper limit) or ECG results, or a clinically significant abnormal outcome at the physical examination at the screening visit;
* have any untreated or uncompensated clinically significant endocrine

disorder;

* have a MINI diagnosis of alcohol and/or drug dependence;
* have a confirmed positive result on the drug screening test for any illicit drug, except cannabis, at Screening;
* be using hormone replacement therapy at Screening;
* have required concomitant treatment with corticosteroids, like

dexamethasone, prednisone or cortisol (topical use is allowed);

* be diagnosed with Cushing's disease;
* be women of childbearing potential without adequate contraception;
* be women with a positive pregnancy test at Screening or Baseline, or

breastfeeding mothers;

* be males with a current diagnosis of prostate hypertrophia or past history (less than 3 months) of symptoms of prostate hypertrophia.
* be currently treated with clozapine (per Amendment III);
* be currently treated with systemic or topical ketaconazole.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2004-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
PANSS positive symptoms subscale. | 6 weeks

SECONDARY OUTCOMES:
Ham-D17, CGI, Cognition, spermatogenesis | 6 weeks